CLINICAL TRIAL: NCT04549701
Title: Inferior Vena CAVA and Lung UltraSound-guided Therapy in Acute Heart Failure: a Randomized Controlled Pilot Trial (CAVAL US-AHF Study)
Brief Title: Inferior Vena CAVA and Lung UltraSound-guided Therapy in Acute Heart Failure
Acronym: CAVAL US-AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Cardiovascular de Buenos Aires (Other)
Responsible Party: Principal Investigator, Lucrecia Maria Burgos, Principal investigator, Instituto Cardiovascular de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 090920
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Acute Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: CAVAL US will be performed on all patients, and patients will be blinded to the assigned group.
  The treating medical team will be blind to the CAVAL US results of the control group.
  Independent clinicians adjudicating 90-day events will not participate in patient follow-up, and will be blind to the assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAVAL US group (Experimental): Patients assigned to this group will receive a daily CAVAL US exam guided decongestive therapy accessible to the treating medical team, in addition to standard care. Diuretic titration: There will not be a specific treatment protocol, but clinicians will be encouraged to tailor treatment, particularly with the use of diuretics, according to the number of B-lines and dilation in the IVC. The therapeutic objective will be discharge patients normal CAVAL US, with relief of congestive signs and symptoms of HF, without electrocardiographic or laboratory alterations that contraindicate discharge.
  Interventions: Other: CAVAL US-guided Therapy; Other: Standard of care
- Standard of care group (Active Comparator): Patients assigned to this group will receive standard care, and diuretic titration will be based on standard practice (physical examination, symptoms, and laboratory results). The therapeutic objective will be discharge patients with relief of congestive signs and symptoms of HF, without electrocardiographic or laboratory abnormalities that contraindicate discharge.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: CAVAL US-guided Therapy — Patients randomly assigned to this group will receive a daily CAVAL US exam guided decongestive therapy accessible to treating medical team, in addition to the standard care.
  Arms: CAVAL US group
Other: Standard of care — Standard of care will be provided.

SUMMARY:
Between 25% and 30% of patients hospitalized for acute heart failure (AHF) are readmitted within 90 days after discharge. Mostly due to persistent congestion on discharge. However, as the optimal evaluation of decongestion is not clearly defined, it is necessary to implement new tools to identify subclinical congestion to guide treatment.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalization of 24 hours or greater for decompensated heart failure defined as new-onset of symptoms or worsening of previous symptoms (including orthopnea, progression to FC III-IV, bendopnea or fatigue) or signs of volume overload.

and - Jugular venous distension, hepatojugular reflux, lower extremity edema or signs of pulmonary congestion.

and

* Chest X-ray with signs suggestive of pulmonary congestion. and
* Elevated ´pro-B-type natriuretic peptide (NT-proBNP) levels of 450 pg/mL, 900 pg/mL, and 1800 pg/mL for ages < 50 years, 50 to 75 years, and > 75 years, respectively, within 24 hours of admission (53,54).

and

- Sufficient ultrasound visualization to assess IVC and lungs.

Exclusion Criteria:

* Not willing to participate.
* Life expectancy of less than 6 months.
* Uninterpretable lung or inferior vena cava ultrasound.
* Transfer to another hospital before hospital discharge.
* SBP < 90 mm Hg.
* Chronic kidney disease (creatinine clearance <30 mL/min calculated with the MDRD equation or hemodialysis).
* Requirement for invasive or noninvasive ventilator support.
* Pregnancy.
* Low cardiac output syndrome/cardiogenic shock.
* Death during index hospitalization.
* Acute coronary syndrome, myocardial revascularization or heart valve replacement within the previous 3 months.
* Being on heart transplant waiting list.
* Cardiac resynchronization therapy device implanted within the previous 3 months.
* Severe tricuspid valve regurgitation.
* Heart failure secondary to causes amenable to invasive correction: cardiac surgery, percutaneous interventions or pacemaker implantation.
* Heart failure secondary to significant arrhythmias (advanced atrioventricular block or sinus arrest, sustained ventricular tachycardia or any sustained arrhythmia other than atrial fibrillation causing hemodynamic instability according to the discretion of the treating physician).
* Heart failure secondary to severe systemic infection
* Severe psychiatric illness
* Palliative care
* SARS-CoV-2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Subclinical congestion at discharge | Discharge

SECONDARY OUTCOMES:
Readmission for heart failure, unplanned visit for worsening HF, or death. | 90 days
  Readmission for heart failure: unscheduled urgent hospital visit and stay longer than 24 hours, requiring medical interventions.
  Mortality: death of the patient. Unplanned visit for worsening heart failure: unscheduled visit to the emergency department that led to an increase in oral / intravenous therapy, stay less than 24 hours.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires, Buenos Aires City
  - Instituto Cardiovascular de Buenos Aires, Buenos Aires, Buenos Aires F.D.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burgos LM, Baro Vila R, Goyeneche A, Munoz F, Spaccavento A, Fasan MA, Ballari F, Vivas M, Riznyk L, Ghibaudo S, Trivi M, Ronderos R, Costabel JP, Botto F, Diez M; CAVAL US-AHF group. Design and rationale of the inferior vena CAVA and Lung UltraSound-guided therapy in Acute Heart Failure (CAVAL US-AHF Study): a randomised controlled trial. Open Heart. 2022 Nov;9(2):e002105. doi: 10.1136/openhrt-2022-002105. PMID 36344108